CLINICAL TRIAL: NCT02380105
Title: Effectiveness of a Counseling Program for TMD Treatment
Brief Title: Effectiveness of a Counseling Program for Temporomandibular Disorders (TMD) Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Rodrigo Falcão Carvalho Porto de Freitas, de Freitas, Universidade Federal do Rio Grande do Norte
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200/11-P CEP/UFRN
Record Dates: First submitted 2014-11-14; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling Group (Experimental): Patients allocated to the counseling group (Group I) were informed about possible etiological factors and educated to not overload the temporomandibular joint and masticatory muscles. Techniques to relieve pain and tension were taught to correct postural habits, food and sleep irregularities. The patients received written instructions, as a way of reinforcing the information provided during the initial consultation. In subsequent returns at 7, 15, 30 and 60 days of follow-up, the instructions were given again and patients were asked whether they had detected any habits related to the initiation and maintenance of painful symptoms of TMD, as a way to further highlight the association between the presence of these harmful behaviors and the worsening signs and symptoms of TMD.
  Interventions: Behavioral: Counseling
- Splint Group (Active Comparator): Patients allocated to the splint group (Group II) were treated using interocclusal appliances, according to the following protocol: At baseline, an anterior bite plate (front-plateau) was made from acrylic resin that was placed in the maxillary arch to include the the canine to canine region and promote the disocclusion of the posterior teeth. Patients were instructed to use the device for 24 hours, interspersed with rests of equal length during the first week. After 7 days, the device was removed. A hard splint was then made. At 30 days of follow-up, the splint was fitted and the patients were also asked to use it when they were sleeping.
  Interventions: Device: Interocclusal Appliances

INTERVENTIONS:
Behavioral: Counseling — Patients were informed of their condition and possible etiological factors contributing to the pathology. They were also educated about the postural rest position of the mandible and instructed to perform bilateral chewing and not overload the temporomandibular joint and masticatory muscles. Techniques to relieve pain and tension were taught to correct postural habits, food and sleep irregularities. The patients received written instructions for future reference, as a way of reinforcing the information provided during the initial consultation.
  Arms: Counseling Group
Device: Interocclusal Appliances — Patients were treated using interocclusal appliances
  Arms: Splint Group

SUMMARY:
This study aims to evaluate the effectiveness of counseling on pain, function and well-fare outcomes for the management of patients with temporomandibular disorder (TMD).

DETAILED DESCRIPTION:
In this study, 51 patients were allocated to one of the research groups. In Group I, it was instituted counseling therapy. For Group II was conducted treatment as usual with occlusal splint. Patients were followed for returns at 7, 15, 30 and 60 days after baseline. At baseline, all patients were examined and assessed Research Diagnostic Criteria/Temporomandibular Disorder (RDC/TMD form). In addition, the patients were referred for specific treatment according to the group to which belonged. In each session, patients were also surveyed about pain intensity using a Numeric Scale. To analyze the impact of pain on quality of life, Oral Health Impact Profile (OHIP-14) questionnaire was used.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals
* Positive diagnosis of TMD according to RDC/TMD
* Presence of pain in the orofacial region persisting for at least a week of at least moderate intensity, according to the Numeric Scale of pain

Exclusion Criteria:

* TMD treatment for ongoing pain
* Presence of pulpal or periodontal disease
* Orthodontic treatment in progress
* Daily use of analgesics, antidepressants or muscle relaxants
* History of radiotherapy to the head and neck, or any adverse systemic condition that may favor presentation of symptoms involved

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pain as measured by Visual Analogue Scale (VAS) | Baseline, 7, 15, 30, 60 days
  Visual Analogue Scale

SECONDARY OUTCOMES:
Quality of life measured by Oral Health Impact Profile (OHIP) | Baseline, 7, 15, 30, 60 days
  Oral Health Impact Profile
Functional Evaluation measured by TemporoMandibular Index (TMI) | Baseline, 7, 15, 30, 60 days
  Temporomandibular Index